CLINICAL TRIAL: NCT01817764
Title: DB2114930: A Randomized, Multi-center, Double-blind, Double-dummy, Parallel Group Study to Evaluate the Efficacy and Safety of Umeclidinium/Vilanterol Compared With Fluticasone Propionate/Salmeterol Over 12 Weeks in Subjects With COPD
Brief Title: A Study to Compare the Efficacy and Safety of Umeclidinium/Vilanterol and Fluticasone Propionate/Salmeterol in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114930
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: umeclidinium bromide (UMEC); vilanterol (VI); salmeterol (SAL); fluticasone propionate (FP); Novel Dry Powder Inhaler (NDPI); Chronic obstructive pulmonary disease; GW642444; GSK573719; lung function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; vilanterol; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium/vilanterol Arm (Experimental): The subjects will receive UMEC/VI 62.5/25 mcg, administered as one inhalation once-daily in the morning via the NDPI and placebo administered as one inhalation each morning and evening via ACCUHALER/DISKUS
  Interventions: Drug: Umeclidinium/vilanterol; Drug: Placebo
- Fluticasone propionate/salmeterol Arm (Active Comparator): The subjects will receive FSC 250/50 mcg, administered as one inhalation each morning and evening via ACCUHALER/DISKUS and placebo administered once-daily in the morning via NDPI
  Interventions: Drug: Fluticasone propionate/salmeterol; Drug: Placebo

INTERVENTIONS:
Drug: Umeclidinium/vilanterol — Dry white powder delivered via NDPI (2 strips with 30 blisters each, first containing UMEC 62.5 mcg per blister and second containing VI 25 mcg per blister), administered as one inhalation of UMEC/VI 62.5/25 mcg once-daily in the morning
  Arms: Umeclidinium/vilanterol Arm
Drug: Fluticasone propionate/salmeterol — Dry white powder delivered via ACCUHALER/DISKUS (1 strip with 60 blisters, containing 250 mcg fluticasone propionate and 50 mcg salmeterol per blister), administered as one inhalation of FSC 250/50 mcg each morning and evening
  Arms: Fluticasone propionate/salmeterol Arm
Drug: Placebo — Placebo will be administered via ACCUHALER/DISKUS or NDPI. Dry white powder administered as one inhalation each morning and evening via ACCUHALER/DISKUS (1 strip with 60 blisters containing placebo) OR once-daily in the morning via NDPI (2 strips with 30 blisters each, containing placebo)

SUMMARY:
This is a multicenter, randomized, double-blind, double-dummy, parallel group study. The purpose of this study is to compare the efficacy and safety of umeclidinium/vilanterol (UMEC/VI) and fluticasone propionate/salmeterol (FSC) in subjects with COPD. Subjects who meet the eligibility criteria at Screening will complete a 7 to 14 day Run-in period. At the end of the run-in period, approximately 710 eligible subjects will be equally randomized (to complete at least 568 evaluable subjects) to one of the 2 treatment groups for 12 weeks: 1. UMEC/VI 62.5/25 micrograms (mcg) administered as one inhalation once-daily in the morning via the Novel dry powder inhaler (NDPI) + placebo administered as one inhalation each morning and evening via single multidose powdered inhaler (ACCUHALER/DISKUS) or 2. FSC 250/50 mcg administered as one inhalation each morning and evening via ACCUHALER/DISKUS + placebo administered once-daily in the morning via NDPI. A safety Follow-up assessment will be conducted approximately 7 days after the end of the study treatment (Early Withdrawal, if applicable). The total duration of subject participation will be approximately 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient
* A signed and dated written informed consent prior to study participation
* Male or female subjects, 40 years of age or older at Visit 1
* A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). - A female is eligible to enter and participate in the study if she is of: Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods as listed in the protocol used consistently and correctly.
* An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society as follows: Chronic obstructive pulmonary disease is a preventable and treatable disease state characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences
* Smoking history: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years (number of pack years = [number of cigarettes per day/20] x number of years smoked [e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years]). Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack year history
* Severity of disease: A pre and post-salbutamol FEV1/Forced Vital Capacity (FVC) ratio of <0.70 and a post-salbutamol FEV1 of >=30% and <=70% of predicted normal values calculated using National Health and Nutrition Examination Survey (NHANES) III reference equations at Visit 1
* Dyspnea: A score of >=2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study
* A current diagnosis of asthma
* Other Respiratory Disorders: Known α-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject, who, in the opinion of the investigator, has any other significant respiratory condition in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Inactive tuberculosis in more than one lobe is exclusionary. Allergic rhinitis is not exclusionary
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, corticosteroid, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic
* Hospitalization for pneumonia within 12 weeks prior to Visit 1
* History of COPD Exacerbation: A documented history of at least one COPD exacerbation in the 12 months prior to Visit 1 that required either oral corticosteroids, antibiotics, and/or hospitalization. Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnea, sputum volume, or sputum purulence
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1)
* 12-Lead Electrocardiogram (ECG): An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility.
* Medication Prior to Spirometry: Unable to withhold salbutamol for the 4 hour period required prior to spirometry testing at each study visit
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids - 12 weeks, Systemic, oral or parenteral corticosteroids - 6 weeks, Antibiotics (for lower respiratory tract infection) - 6 weeks, Cytochrome P450 3A4 strong inhibitors - 6 weeks, Herbal medications potentially containing oral or systemic steroids - 6 weeks, Inhaled corticosteroids (ICS) - 30 days, Long-acting beta2-agonist (LABA)/ICS combination products - 30 days, Phosphodiesterase 4 (PDE4) inhibitors (e.g., roflumilast) - 14 days, Inhaled long-acting anticholinergics - 7 days, Theophyllines - 48 hours, Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton) - 48 hours, Oral beta2-agonists Long-acting-48 hours/Short-acting - 12 hours, Inhaled long acting beta2-agonists (LABA, e.g., salmeterol, formoterol, indacaterol) - 48 hours, Inhaled sodium cromoglycate or nedocromil sodium - 24 hours, Inhaled short acting beta2-agonists - 4 hours, Inhaled short-acting anticholinergics - 4 hours, Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products - 4 hours, Any other investigational medication - 30 days or within 5 drug half-lives (whichever is longer)
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not exclusionary
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1
* Affiliation with Investigator Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator
* Inability to read: A subject will not be eligible for the study if in the opinion of the investigator the subject cannot read

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2013-03-01; Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (9):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
- Argentina (5):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (5):
  - GSK Investigational Site, Quillota, Región de Valparaíso
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Viña del Mar
- Greece (5):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari / Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Rethymnon, Crete
  - GSK Investigational Site, Thessaloniki
- GSK Investigational Site, Lima, Lima Province, Peru
- Romania (8):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Ukraine (8):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Yalta

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Donohue JF, Worsley S, Zhu CQ, Hardaker L, Church A. Improvements in lung function with umeclidinium/vilanterol versus fluticasone propionate/salmeterol in patients with moderate-to-severe COPD and infrequent exacerbations. Respir Med. 2015 Jul;109(7):870-81. doi: 10.1016/j.rmed.2015.04.018. Epub 2015 May 8. PMID 26006754
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114930 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114930 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114930 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114930 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114930 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114930 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114930 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 707 participants, representing the enrolled participants, were randomized to study treatment. Of these, 706 comprised the Intent-to-Treat Population (participants randomized to treatment who received >=1 dose of randomized study medication in the treatment period).
Groups:
- UMEC/VI 62.5/25 µg QD: Participants were randomized to umeclidinium bromide/vilanterol (UMEC/VI) 62.5/25 micrograms (µg) once-daily (QD) treatment in the morning via a dry powder inhaler (DPI) and placebo in the morning and evening via a separate DPI.
- FSC 250/50 µg BID: Participants were randomized to fluticasone propionate/salmeterol (FSC) 250/50 µg twice-daily (BID) treatment in the morning and evening via a DPI and placebo in the morning via a separate DPI.
Period: Overall Study
Arm/Group | UMEC/VI 62.5/25 µg QD | FSC 250/50 µg BID
Started | 353 | 353
Completed | 319 | 315
Not Completed | 34 | 38
Not completed — Adverse Event | 7 | 10
Not completed — Lack of Efficacy | 9 | 7
Not completed — Protocol Violation | 7 | 5
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UMEC/VI 62.5/25 µg QD | FSC 250/50 µg BID | Total
Number analyzed (Participants) | 353 | 353 | 706
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (9.05) | 63.0 (8.91) | 62.8 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 109 | 209
  Male | 253 | 244 | 497
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 4 | 3 | 7
  American Indian or Alaska Native | 5 | 5 | 10
  Asian - East Asian Heritage | 1 | 1 | 2
  Asian - Japanese Heritage | 2 | 1 | 3
  White - Arabic/North African Heritage | 0 | 1 | 1
  White - White/Caucasian/European | 341 | 342 | 683

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Weighted-mean Serial FEV1 on Treatment Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Weighted mean is calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5 and 15 minutes and 1, 3, 6, 9, 12 (pre-evening dose), 13, 15, 18, 23, and 24 hours after the morning dose. Change from Baseline was calculated as the value at Day 84 minus the value at Baseline. Analysis was performed using an analysis of covariance of treatment, Baseline (mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1), and smoking status. par.=participants.
Time Frame: Baseline and Day 84
Population: Intent-to-Treat (ITT) Population: all par. randomized to treatment who received >=1 dose of randomized study medication in the treatment period. Only par. with analyzable data at the indicated time point were assessed, but all par. without missing covariate information and with >=1 post-Baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 µg QD | FSC 250/50 µg BID
Number analyzed (Participants) | 315 | 310
Liters | 0.165 (0.0130) | 0.091 (0.0131)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 µg QD vs FSC 250/50 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 0.074, 95% CI 2-sided [0.038 to 0.110]

2. Secondary Outcome: Change From Baseline in Trough FEV1 on Day 85
Description: Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained 23 and 24 hours after morning dosing/11 and 12 hours after evening dosing on Day 84. Change from Baseline is calculated as the Day 85 value minus the Baseline value. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1), smoking status, day, and day by Baseline and day by treatment interactions.
Time Frame: Baseline and Day 85
Population: ITT Population. Only those participants with analyzable data at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 µg QD | FSC 250/50 µg BID
Number analyzed (Participants) | 317 | 312
Liters | 0.154 (0.0133) | 0.072 (0.0134)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the follow-up contact (up to 13 weeks).
Description: On-treatment SAEs and non-serious AEs were reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study drug in the treatment period.
Arm/Group | UMEC/VI 62.5/25 µg QD | FSC 250/50 µg BID
Serious Adverse Events (participants affected / at risk) | 6/353 | 10/353
Other Adverse Events (participants affected / at risk) | 38/353 | 25/353
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 µg QD (N=353) | FSC 250/50 µg BID (N=353)
Pneumonia (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 0 | 1
Burn infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 µg QD (N=353) | FSC 250/50 µg BID (N=353)
Headache (Nervous system disorders) | 23 | 17
Nasopharyngitis (Infections and infestations) | 16 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.